CLINICAL TRIAL: NCT00401999
Title: OPRM1 A118G SNP, Alcohol Response, and Striatal Dopamine
Status: Completed | Type: Observational
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070026; 07-AA-0026
Record Dates: First submitted 2006-11-18; First posted 2006-11-22 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-01-28

CONDITIONS: Alcoholism
Keywords: PET; C-11 Raclopride; Dopamine; OPRM1; Alcohol; Healthy Volunteer; HV
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will examine the relationship between variations in a gene called OPRM1 and the response to alcohol. The OPRM1 (Mu-opioid Receptor-1) gene helps regulate brain pathways involved in experiencing pleasure. Brain pathways use a chemical called dopamine. Different forms of the OPRM1 gene may lead to differences in how dopamine is released and subsequently to differences in a person's response to alcohol.

Healthy non-smokers between 21 and 45 years of age may be eligible for this study. Candidates are screened with a medical and psychiatric history and physical examination, blood and urine tests, and breathalyzer (breath alcohol test). A blood test is also done to determine the variant of OPRM1 gene.

Participants undergo the following procedures in three study sessions:

Session 1

" Breathalyzer test, urine test for illicit drugs and pregnancy test for women who can become pregnant.

" Insertion of catheters (plastic tubes) into a vein in one arm for infusing alcohol and into the other arm for drawing blood samples.

" Completion of questionnaires on how intoxicated the subject feels.

" Blood draw for research studies.

" Eye movement test (a visor with a digital camera tracks the subject's eye movements while he or she watches lights on a computer screen).

" 45-minute alcohol infusion (up to 0,08 grams per deciliter - a level considered in most states as driving under the influence of alcohol).

" Repeat breathalyzer, questionnaires, eye movement test and blood draw every 15 minutes during the infusion and again after the infusion is complete.

" Subjects remain in the clinic until their blood alcohol content falls below 0.02 g/dL, determined by a breathalyzer test done every 15 minutes. Subjects can usually return home about 3 to 4 hours after the alcohol infusion stops.

Sessions 2 and 3

The procedure is the same as for session 1, except subjects receive an infusion of alcohol one session and an infusion of saline (salt water) the other. Also, subjects undergo positron emission tomography (PET) scanning during the infusions. For this test, the subject lies on a bed that slides in and out of a doughnut-shaped scanner. A custom-molded mask is used to support the head and prevent it from moving during the scanning. A small amount of radioactive substance called C-11 raclopride is injected through one of the catheters to trace brain dopamine activity.

...

DETAILED DESCRIPTION:
Objectives:

Reinforcing properties of alcohol are in part mediated through endogenous opioids. Mesolimbic dopamine (DA) release is a key signal for drug reward, and endogenous opioids are thought to exert their effects by modulating the activity of this system. A functional mu-opioid receptor (OPRM1) A118G single nucleotide polymorphism (SNP) alters the affinity of the mu-opioid receptor for its endogenous ligand, is in some studies associated with increased risk for alcohol and heroin addiction, and confers differential pain sensitivity and subjective responses to alcohol. This prompts the question whether the differential subjective response to alcohol observed as a function of the OPRM1 A118G genotype reflects differential activation of the mesolimbic DA release. The objective of this study is to examine the role of the A118G OPRM1 polymorphism for responses to a highly standardized intravenous alcohol challenge, with regard to psycho-physiological variables measured in the laboratory, and for brain dopamine release measured by 11C raclopride PET.

Study Population:

We will screen healthy participants from the general population to obtain samples of two groups of subjects: 1) persons homozygous for the major 118A allele (118AA genotype); 2) persons carrying one or two copies of the variant 118G allele (118AG or 118GG genotype, hereafter called 118GX).

Design and Outcome Measures:

We will compare the response of these groups to a standardized alcohol challenge using the procedure in place for NIAAA protocols 03-AA-0283 Influence of Age and Gender on Alcohol Metabolism and Acute Responses and 04-AA-0060 The Effect of Ethanol on Cerebral Blood Flow as Measured by Functional Magnetic Resonance Imaging and the Development of Conditioned Response to Ethanol Administration . Participants will be given a standardized IV infusion of an alcohol solution infused to achieve and maintain a target blood alcohol level of 80 mg%. Pre and post infusion measures will be made in two areas: 1) subjective response as measured by standardized questionnaires, and 2) measures of physiologic response, to include saccadic eye movements and blood chemistries. We hypothesize that 118GX subjects will have significantly higher subjective response to alcohol challenge than 118AA subjects. We will then repeat the alcohol infusion procedure in all participants twice in the PET scanner, infusing alcohol or saline, and assess displacement of 11C raclopride, a positron emitter labeled ligand which binds preferentially to D2 receptors. We hypothesize that 118GX subjects will have more 11C raclopride displacement after alcohol infusion relative to placebo, indicating greater amounts of dopamine release.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Male and female participants between 21-45 years of age.
  2. Good health as determined by medical history, physical exam, EKG and lab tests.
  3. Social drinkers consuming less than 20 alcoholic beverages per week, on average, having normal liver enzymes and not seeking treatment for alcohol-related problems.
  4. Current non-smokers who have never smoked or quit at least a year prior to enrolling in the study.
  5. Females will have normal menstrual cycles and will be tested during the follicular phase of their cycle (within 15 days of offset of menses) and must have a negative urine pregnancy (hCG) test at the start of each study session.
  6. An equal number of final participants will be of OPRM1 118 A/A vs. 118A/G or 118G/G genotype.

EXCLUSION CRITERIA:

1. Current or prior history of any significant disease, including cardiovascular, respiratory, gastrointestinal, hepatic, renal, endocrine, or reproductive disorders, or a positive hepatitis or HIV test at screening.
2. Current Axis-I psychiatric illness.
3. Current or prior history of any alcohol or drug dependence, as well as non-drinkers (alcohol-naive individuals or current abstainers).
4. Positive result on urine screen for illicit drugs.
5. Nursing, pregnancy or intention to become pregnant for women. Female participants will undergo a clinical interview and a urine beta-hCG test to ensure they are not pregnant. If it is not possible to document non-pregnancy, the study will not be performed.
6. Inability to undergo an MRI scan of the brain due to claustrophobia or anxiety when confined to small spaces such as the magnet bore, or due to the presence of metallic implants.
7. Use of prescription or OTC medications known to interact with alcohol within 2 weeks of the study. These include, but may not be limited to: isosorbide, nitroglycerine, benzodiazepines, warfarin, anti-depressants such as amitriptyline, clomipramine and nefazodone, anti-diabetes medications such as glyburide, metformin and tolbutamide, H2-antagonists for heartburn such as cimetidine and ranitidine, muscle relaxants, anti-epileptics including phenytoin and phenobarbital codeine, and narcotics including darvocet, percocet and hydrocodone. Drugs known to inhibit or induce enzymes that metabolize alcohol should not be used for 4 weeks prior to the study. These include chlorzoxazone, isoniazid, metronidazole and disulfiram. Cough-and-cold preparations which contain anti-histamines, pain medicines and anti-inflammatories such as aspirin, ibuprofen, acetaminophen, celecoxib and naproxen, should be withheld for at least 72 hours prior to each study session.
8. Self-reported history of flushing upon intake of alcohol.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2006-11-16; Study Completion 2011-01-28

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kreek MJ, LaForge KS, Butelman E. Pharmacotherapy of addictions. Nat Rev Drug Discov. 2002 Sep;1(9):710-26. doi: 10.1038/nrd897. PMID 12209151
- [Background] Contet C, Kieffer BL, Befort K. Mu opioid receptor: a gateway to drug addiction. Curr Opin Neurobiol. 2004 Jun;14(3):370-8. doi: 10.1016/j.conb.2004.05.005. PMID 15194118
- [Background] Roberts AJ, McDonald JS, Heyser CJ, Kieffer BL, Matthes HW, Koob GF, Gold LH. mu-Opioid receptor knockout mice do not self-administer alcohol. J Pharmacol Exp Ther. 2000 Jun;293(3):1002-8. PMID 10869404